CLINICAL TRIAL: NCT05719103
Title: Changes in Lung Aeration and Inspiratory Effort During High-Flow Nasal Oxygen and Non-Invasive Mechanical Ventilation With and Without Awake Prone
Brief Title: Changes in Lung Aeration and Inspiratory Effort With and Without Awake Prone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: APP-HF-NIV
Record Dates: First submitted 2023-01-16; First posted 2023-02-08 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Respiratory Distress Syndrome; Ventilation Therapy; Complications
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- HFNC SP (Active Comparator): HFNC flow at 60 L/min or maximum tolerable flow at supine position
  Interventions: Behavioral: With and Without Awake Prone Positioning
- HFNC PP (Active Comparator): HFNC flow at 60 L/min or maximum tolerable flow at prone position
  Interventions: Behavioral: With and Without Awake Prone Positioning
- NIV SP (Active Comparator): CPAP with full face mask at 10 cmH2O at supine position
  Interventions: Behavioral: With and Without Awake Prone Positioning
- NIV PP (Active Comparator): CPAP with full face mask at 10 cmH2O at prone position
  Interventions: Behavioral: With and Without Awake Prone Positioning
- MC SP (Placebo Comparator): Mask oxygen at supine position
  Interventions: Behavioral: With and Without Awake Prone Positioning
- MC PP (Placebo Comparator): Mask oxygen at prone position
  Interventions: Behavioral: With and Without Awake Prone Positioning

INTERVENTIONS:
Behavioral: With and Without Awake Prone Positioning — 1. HFNC flow at 60 L/min or maximum tolerable flow at supine position
  2. HFNC flow at 60 L/min or maximum tolerable flow at prone position
  3. CPAP with full face mask at 10 cmH2O at supine position
  4. CPAP with full face mask at 10 cmH2O at prone position
  5. MC at supine position
  6. MC at prone position
  Other Names: HFNC and NIV

SUMMARY:
The investigators aimed to investigate the ventilation homogeneity and transpulmonary pressure during treatments of High-flow nasal cannula(HFNC) and (CPAP) on supine and prone position for COVID-19 or non-COVID-19 patients with acute hypoxemic respiratory failure (AHRF).

DETAILED DESCRIPTION:
Awake prone positioning (APP) for non-intubated patients has been reported to improve oxygenation for patients with acute hypoxemic respiratory failure (AHRF),particularly for patients with COVID-19 induced AHRF, APP has been shown to decrease the need of intubation.Similarly, APP with helmet continuous positive airway pressure (CPAP) enables a reduction in the work of breathing and an improvement in oxygenation and sensation of dyspnea in COVID-19-associated acute respiratory distress syndrome (ARDS). Moreover, among intubated patients with ARDS assessed by electro-impedance tomography (EIT), prone positioning was found to reduce alveolar overdistention and collapse, resulting in improvement of ventilation homogeneity.However, the effects of APP on the ventilation homogeneity and work of breathing for non-COVID-19 patients with AHRF remain unknown.

High-flow nasal cannula (HFNC) has been proven to improve oxygenation and reduce intubation rate for patients with AHRF in multiple meta-analyses,and has been recommended to treat AHRF in several recently published guidelines.CPAP provides consistent level of positive end-expiratory pressure (PEEP), in comparison to variable level of PEEP generated by HFNC, thus CPAP was reported to have greater improvement of oxygenation than HFNC in 20 patients with AHRF, more importantly, they found that among patients who avoided intubation, the extent of oxygenation improvement was greater with HFNC+APP than with NIV+APP, in contrast, for patients who were intubated, the extent of oxygenation improvement was greater with NIV+APP than with HFNC+APP.This raised the concerns of the self-inflicted lung injury (SILI) generated by heterogenous aeration and large swings of transpulmonary pressure. Thus, the investigators aimed to investigate the ventilation homogeneity and transpulmonary pressure during treatments of HFNC and CPAP on supine and prone.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18-90 years) who have acute hypoxemic respiratory failure, requiring FIO2 > 0.4 to maintain SpO2 at 90-95% during HFNC at 50 L/min

Exclusion Criteria:

* patients who need immediate intubation; refuse to participate in the study; unable to communicate; have contraindication to place the esophageal catheter; unable to use EIT, such as open-chest surgery with chest tube placement; have contraindication for prone positioning, including pregnant, post-abdomen surgery within a week; hypercapnic respiratory failure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The differences in lung homogeneity during HFNC | 30 minutes
  The differences in lung homogeneity (global inhomogeneity index) during HFNC therapy at 60 L/min or maximum tolerable flow at supine and awake prone position
The differences in lung homogeneity during CPAP | 30 minutes
  The differences in lung homogeneity (global inhomogeneity index) during CPAP with full face mask at 8 cmH2O at supine and awake prone position

SECONDARY OUTCOMES:
patient' comfort scores | 30 minutes
  during HFNC and CPAP treatment at supine and prone position, patient' comfort scores
work of breathing | 30 minutes
  the differences in WOB during HFNC therapy at 60 L/min or maximum tolerable flow at supine and awake prone position

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhong, MD, phD, Study Chair — Fudan University
Locations (1):
- Zhongshan hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No